CLINICAL TRIAL: NCT04512261
Title: TOPAZ: Single Arm, Open Label Phase 1b/2 Study of Tucatinib in COmbination With Pembrolizumab And TrastuZumab in Patients With HER2-Positive Breast Cancer Brain Metastases
Brief Title: TOPAZ: Tucatinib in COmbination With Pembrolizumab And TrastuZumab in Patients With HER2-Positive Breast Cancer Brain Metastases
Acronym: TOPAZ
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to change in treatment landscape for HER2+ metastatic breast cancer.
Sponsor: Reva Basho (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Reva Basho, Assistant Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2019-21-Basho-TOPAZ
Record Dates: First submitted 2020-07-28; First posted 2020-08-13 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Brain Metastases; HER2-positive Breast Cancer; CNS Disease
Keywords: tucatinib; pembrolizumab; trastuzumab
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Central Nervous System Diseases | interventions — tucatinib; pembrolizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib + Pembrolizumab + Trastuzumab (Experimental): Patients will receive a combination therapy of tucatinib with pembrolizumab and trastuzumab during the treatment period until progression, treatment intolerance, or patient withdrawal from study. Tucatinib and pembrolizumab are administered as experimental use while trastuzumab is administered per standard use. Patients are expected to be on treatment for at least 12 weeks.
  Interventions: Drug: Tucatinib; Drug: Pembrolizumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Tucatinib — Initial dosage of trial treatment for tucatinib will be given as 300 mg (dispensed as 2 x 150 mg tablets) orally twice a day for Days 1 - 21 of each 3-week cycle during the treatment period.
  Other Names: Tukysa
Drug: Pembrolizumab — Initial dosage of trial treatment for pembrolizumab will be given as 200 mg by intravenous infusion every 3 weeks on Day 1 of each 3-week cycle during the treatment period. Pembrolizumab will be administered for a maximum of 35 doses.
  Other Names: Keytruda
Drug: Trastuzumab — Initial dosage of trial treatment for trastuzumab will be given as 8 mg/kg by intravenous (IV) infusion once on Day 1 of Cycle 1, and 6 mg/kg by IV every 3 weeks on Day 1 of each 3-week cycle starting on Cycle 2 during the treatment period.
  Other Names: Herceptin

SUMMARY:
This is a single arm, open label trial to assess the safety and efficacy of tucatinib in combination with pembrolizumab and trastuzumab for the treatment of HER2+ breast cancer brain metastases (BCBM). A total of 33 patients with untreated or previously treated and progressing HER2+ BCBM not requiring urgent central nervous system (CNS)-directed therapy will be enrolled. The study will determine the recommended dose of tucatinib in this combination and assess the efficacy of this combination in controlling CNS disease in patients with HER2+ BCBM.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. ECOG performance status of 0-2.
3. HER2+ (as defined by ASCO/CAP clinical practice guideline) metastatic breast cancer.
4. Untreated or previously treated and progressing CNS disease.
5. Measurable CNS metastases.
6. Must be able to undergo MRI of the brain.
7. Adequate organ function.

Exclusion Criteria:

1. Any indication for immediate CNS-directed therapy.
2. History of generalized or complex partial seizures.
3. Any other manifestation of neurologic progression that in the opinion of the treating physician is due to brain metastases.
4. Leptomeningeal disease.
5. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
6. Prior therapy with tucatinib.
7. Active autoimmune disease that has required systemic treatment in excess of prednisone 10mg daily or equivalent in the past 2 years.

Complete inclusion/exclusion criteria are detailed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
24-week CNS disease control rate (DCR) | 24 weeks
  Percentage of patients who experience objective tumor response [ partial response (PR) or complete response (CR) ] or stable disease as assessed by investigator per RANO-BM reads on protocol-specified MRIs of the brain.
Recommended dose of tucatinib in combination with pembrolizumab and trastuzumab | 24 weeks

SECONDARY OUTCOMES:
CNS objective response rate (ORR) | From baseline until the date of first documented progression or study discontinuation. Assessed up to 2 years.
  Proportion of participants with confirmed CR or PR per RANO-BM Criteria
Systemic ORR | From baseline until the date of first documented progression or study discontinuation. Assessed up to 2 years.
  Proportion of participants with confirmed CR or PR per RECIST v.1.1
Progression-free survival (PFS) | From baseline to first documentation of true progression or symptomatic deterioration, or death due to any cause. Assessed up to 2 years.
  From date of registration to date of first documentation of true progression or symptomatic deterioration (as defined above), or death due to any cause. Patients last known to be alive and progression free are censored at date of last assessment. PFS will be assessed in the CNS and systemically.
Overall Survival (OS) | From baseline until death or 3 years, whichever occurs first.
  From date of registration to date of death due to any cause. Patient's last known to be alive are censored at date of last contact.
Toxicity profile of tucatinib, pembrolizumab, and trastuzumab co-administration | From first dose of study treatment until 30 days after the last dose of study treatment.
  Number of adverse events as assessed per CTCAE v.5.

CONTACTS AND LOCATIONS:
Overall Officials: Reva Basho, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States